CLINICAL TRIAL: NCT02126488
Title: Perturbation Training for Fall-risk Reduction Among Older Adults
Brief Title: Effect of Adaptive Training for Balance Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Tanvi Bhatt, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000-0788; R01AG044364 (NIH)
Record Dates: First submitted 2014-04-25; First posted 2014-04-30 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Balance, Postural; Prevention, Accident
Keywords: treadmill training; generalization; retention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- treadmill perturbation (Experimental): treadmill slip perturbation
  Interventions: Behavioral: treadmill slip perturbation
- treadmill placebo (Placebo Comparator): treadmill training placebo
  Interventions: Behavioral: treadmill training placebo
- observation (Sham Comparator): observation training
  Interventions: Behavioral: observation training

INTERVENTIONS:
Behavioral: treadmill slip perturbation — Group A will receive perturbation training on a treadmill with precisely controlled slip-like displacements and then encounter an unannounced novel slip during over-ground walking.
  Arms: treadmill perturbation
Behavioral: treadmill training placebo — An age-matched control group (Group B) will receive only placebo training (on the same treadmill for the same duration but without perturbation) but encounter an identical novel slip during their over-ground walking.
  Arms: treadmill placebo
Behavioral: observation training — An age-matched observation-training group (Group C) will watch a training video and slides. When exposed to an identical novel slip in over-ground walking, they will know where and how the slip is going to occur and how to resist a fall.
  Arms: observation

SUMMARY:
The long-term objective of this research is a prophylactic approach that can reduce the incidence of falls and the resulting injuries among older adults at risk and thus reduce its escalating medical cost. This project explores perturbation training through the use of treadmill device and a motor learning approach, in which experience with slip-like perturbation generated by that treadmill is used to prepare the motor system to develop and then put to use fall-resisting skills outside of training environment (cross-environment transfer). The computer-controlled treadmill is portable, safe and easy to operate, thus conducive for use in clinics or community centers. The study logically builds on and complements the team's previous and current research programs, and will further test that after such a single session, older adults at risk can retain such cross-environment transfer and reduce their likelihood of falls in everyday living for the next 6 to 12 months. Finally, the study will explore that such reduction of falls does not come merely from these persons' familiarity with the training or testing setup, protocol and environments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with no known history of musculoskeletal, neurological, cardiovascular, or pulmonary impairment that may affect their ability to perform the testing procedures will be included.

Exclusion Criteria:

* Ultrasound calcaneus bone mineral density T score < -2.5 (osteoporotic)
* Mini-Mental State exam score < 25 (cognitive impairment)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 308 (Actual)
Dates: Start 2014-06; Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Fall incidence | 1 year

SECONDARY OUTCOMES:
Dynamic stability | 6 months
  The dynamic stability will be evaluated based on the dynamic relationship of motion state (i.e., the combination of position and velocity) between the center of mass and the base of support. It will be calculated as the shortest distance from the instantaneous motion state of the center of mass to the threshold against backward fall. It is a dimensionless variable.

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi Bhatt, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Clinical Gait and Movement Analysis Laboratory, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wang Y, Wang S, Liu X, Lee A, Pai YC, Bhatt T. Can a single session of treadmill-based slip training reduce daily life falls in community-dwelling older adults? A randomized controlled trial. Aging Clin Exp Res. 2022 Jul;34(7):1593-1602. doi: 10.1007/s40520-022-02090-3. Epub 2022 Mar 2. PMID 35237948